CLINICAL TRIAL: NCT06381804
Title: Effect of Shotblocker and Palm Stimulator in Reducing Pain Associated With Intramuscular Injection: A Randomized Controlled Trial
Brief Title: Effect of Shotblocker and Palm Stimulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gulden Basit, Assist. Prof., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24YL9001
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- shotblocker (Experimental): shotblocker
  Interventions: Other: shotblocker
- palm stimulator (Experimental): palm stimulator
  Interventions: Other: palm stimulator
- control (No Intervention): control

INTERVENTIONS:
Other: shotblocker — shotblocker device
  Arms: shotblocker
Other: palm stimulator — palm stimulator
  Arms: palm stimulator

SUMMARY:
This study discusses the advancements in nursing, particularly focusing on intramuscular injections, their complications, and innovative non-pharmacological methods such as the Shotblocker and palm stimulator to reduce pain. These methods, based on the gate control theory, aim to minimize discomfort during injections by applying tactile stimulation, which has proven effective in various studies.

DETAILED DESCRIPTION:
It was planned to examine the effect of shot blocker and palm stimulator use on injection-related pain during intramuscular injection.This study is a randomized controlled, single-blind, parallel group experimental study to be conducted in the emergency department of a State Hospital in Konya, Turkey. The research will be conducted on individuals who will receive intramuscular (IM) injection. Participants will be randomized and divided into Shotblocker, Palm stimulator and control groups. Data collection will run from April 2024 to May 2024 and analyzes will be conducted blinded by an independent statistician. This study aims to evaluate the effects of these techniques on pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,

  * Those who will receive vitamin B injection ordered by physician due to B12 deficiency,
  * Conscious and oriented,
  * Able to understand and speak Turkish,
  * Age range is between 18-65,
  * Having no vision or hearing problems,
  * Pain score of 2 or less when evaluated with a visual analog scale,
  * Able to lie in the right lateral position where injection can be administered,
  * Those who have not had an IM injection into the right ventrogluteal area in the last week,
  * Body mass index is within the normal range (25.0-29.9 kg/m2) according to WHO,
  * Those who have not used any analgesics or muscle relaxants in the last 24 hours,
  * Does not have any problems such as hardness, mass, edema or infection in the area to be injected,
  * According to his own statement, he has no psychiatric diagnosis,

Exclusion Criteria:

* Having pain anywhere in the body,

  * Narcotic type or different analgesic area before application,
  * Pregnant or suspected of pregnancy,
  * Individuals in menstrual period,
  * Receiving chemotherapy and radiotherapy treatment,
  * Those who have migraine, are in the postoperative period, have nerve damage, neuropathy and a vascular disease,
  * Those who have disabilities in grasping their hands,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) pain Scale score | up to 6 weeks
  The Visual analog scale (VAS) score for grading of pain consists of a 10 centimetres (cm) line with 10 mm (0.01 cm) to each point of the scale and two end-points representing no pain and worst possible pain, where 0 = no pain, 1-3 = mild, 4-6 = moderate and 7-10 = severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Gülden Basit, PhD, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No